CLINICAL TRIAL: NCT07076186
Title: Phase II Decentralized Pragmatic Trial of Adjuvant Doxorubicin - Trabectedin Chemotherapy in Uterine Leiomyosarcoma
Brief Title: Phase II Decentralized Pragmatic Trial of Adjuvant Doxorubicin - Trabectedin Chemotherapy in uLMS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0352; NCI-2025-05088 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Uterine Leiomyosarcoma
MeSH Terms: interventions — Trabectedin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase II Single Arm Treatment with Doxorubicin and Trabectedin (Experimental): Participants will receive treatment on an outpatient and standard of care basis
  Interventions: Drug: Trabectedin; Drug: Doxorubicin Hydrochloride

INTERVENTIONS:
Drug: Trabectedin — Given by IV Infusion
Drug: Doxorubicin Hydrochloride — Given by IV Infusion

SUMMARY:
To find out if receiving standard chemotherapy (doxorubicin and trabectedin) can extend the cancer-free survival of patients with Stage 1b/2 uterine leiomyosarcoma who had surgery that fully removed the tumor.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate disease-free survival (DFS) in patients with FIGO stage 1b and 2 uterine leiomyosarcoma receiving adjuvant chemotherapy by standard-of-care doxorubicin and trabectedin for 6 cycles

Secondary Objectives:

To assess overall survival (OS) in patients with FIGO stage 1b and 2 uterine leiomyosarcoma receiving adjuvant chemotherapy by standard-of-care doxorubicin and trabectedin for 6 cycles

* To characterize treatment-related toxicity according to Common Terminology Criteria for Adverse Events (CTCAE), in patients with FIGO stage 1b and 2 uterine leiomyosarcoma receiving adjuvant chemotherapy by standard-of-care doxorubicin and trabectedin for 6 cycles
* To evaluate quality of life (QoL) outcomes using patient-reported measures in patients with FIGO stage 1b and 2 uterine leiomyosarcoma receiving adjuvant chemotherapy by standard-of-care doxorubicin and trabectedin for 6 cycles
* To analyze ctDNA dynamics as a predictor of treatment response and recurrence risk, in patients with FIGO stage 1b and 2 uterine leiomyosarcoma receiving adjuvant chemotherapy by standard-of-care doxorubicin and trabectedin for 6 cycles
* To estimate the incidence of germline genetic alterations in patients with localized uLMS

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed uterine leiomyosarcoma
* Patients must have localized tumors, AJCC stages 1b to 3 according to the AJCC uterine sarcoma staging system (high risk of relapse population)
* Patients must have had complete surgical resection of tumor within 3 months prior to initiation of adjuvant chemotherapy, complete surgical resection includes at least a total hysterectomy
* Patients must have no evidence of residual disease, as proven by CT Chest-Abdomen-Pelvic within 28 days before randomization (exclude potential metastatic patients)
* Patients must have no history of pelvic radiation (hematologic tolerance of chemotherapy is impaired by pelvic radiation)
* No prior chemotherapy for the treatment of the uterine leiomyosarcoma
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of doxorubicin in combination with trabectedin in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤2 (Karnofsky ≥60%,).
* Patients must have adequate organ and marrow function as defined below:
* absolute neutrophil count ≥1,000/mcL
* platelets ≥100,000/mcL
* total bilirubin ≤ institutional upper limit of normal (ULN) (except patients with Gilbert's syndrome, who must have total bilirubin < 3.0 mg/dL)
* AST(SGOT)/ALT(SGPT) ≤2× institutional ULN
* eGFR (using 2021 CKD-EPI) ≥40mL/min/1.73m2
* Albumin > 2.8mg/dL
* CPK ≤2× institutional ULN
* No cardiac dysfunction as proven by LVEF>50%
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to doxorubicin or trabectedin or other agents used in study.
* Patients with uncontrolled intercurrent illness per clinical judgment of the study PI and/or treating physician
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-02 (Estimated); Study Completion 2029-12-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Elise Nassif Haddad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org